CLINICAL TRIAL: NCT05799287
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Telitacicept in Patients With Primary IgA Nephropathy
Brief Title: A Study of Telitacicept for IgA Nephropathy (TELIGAN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C021
Record Dates: First submitted 2023-03-05; First posted 2023-04-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Primary IgA Nephropathy
Keywords: Autoimmune Diseases; Immune System Diseases; IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Autoimmune Diseases; Immune System Diseases | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Subjects will be given Telitacicept 240 mg SC once a week in phase A for a total of 39 doses and once every 2 weeks in phase B for a total of 32 doses.
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Subjects will be given placebo SC once a week in phase A for a total of 39 doses and once every 2 weeks in phase B for a total of 32 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Subcutaneous injection
  Other Names: RC18
  Arms: Telitacicept
Drug: Placebo — Placebo to Telitacicept
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Telitacicept in patients with primary IgA nephropathy at risk of progressing to end-stage renal disease(ESRD), despite maximum tolerated treatment with renin-angiotensin system(RAS) blockade using angiotensin converting enzyme inhibitors (ACEIs) or angiotensin II type I receptor blockers (ARBs).

DETAILED DESCRIPTION:
This study consists of a 5-week screening period, a double-blind treatment period divided into phase A and phase B. Eligible subjects will be randomly assigned in a 1:1 ratio to receive either Telitacicept 240mg or placebo. Subjects will be given subcutaneous injection（SC） Telitacicept or placebo once a week for a total of 39 doses in phase A and once every 2 weeks for a total of 32 doses in phase B.

Primary endpoint of phase A will be measured at week 39. Primary endpoint of phase B will be measured at week 104.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent provided;
2. Male or female aged ≥ 18 years old;
3. IgA nephropathy confirmed by pathological biopsy;
4. During the screening period, UPCR ≥ 0.8 g/g or 24-hour urine protein ≥ 1.0 g/day based on 24-hour urine collection at Visit 1 and/or Visit 2 and at Visit 3;
5. eGFR ≥ 30 mL/min per 1.73 m^2 (using the CKD-EPI);
6. Have been on a treatment regimen including ACEI/ARB for 12 weeks and on a stable use of ACEI/ARB medication at the maximum tolerated dose/maximum allowable dose within 4 weeks prior to randomization. Subjects who use both ACEIs and ARBs will be excluded.

Exclusion Criteria:

1. Subjects with abnormal laboratory tests, including but not limited to the following:

   1. White blood cell count < 1.5×109/L
   2. Neutrophils < 1.0×109/L
   3. Hemoglobin < 85.0 g/L
   4. Platelet count < 80.0×109/L
   5. Total bilirubin >2×ULN
   6. ALT>3×ULN
   7. AST>3×ULN
   8. Alkaline phosphatase>2×ULN
   9. Creatine kinase>5×ULN
   10. IgA<10 mg/dL; or IgG≤400mg/dL；
2. Patients with secondary IgA nephropathy, including but not limited to: Henoch-Schonlein purpura, ankylosing spondylitis, systemic lupus erythematosus, etc.;
3. Patients with other types of glomerular disease such as crescentic glomerulonephritis, minimal change nephropathy with IgA deposition;;
4. Renal transplant;
5. Patients with cirrhosis, as assessed by the investigator;
6. Patients who experienced any of the following cardiovascular and cerebrovascular events within 24 weeks prior to randomization: myocardial infarction, unstable angina, ventricular arrhythmia, NYHA Class II or higher heart failure, stroke, etc.;
7. Sitting position SBP>140 mmHg or DBP>90 mmHg for at least once at 2 visits during the screening period;
8. Patients with poorly controlled type 1 and type 2 diabetes (glycated hemoglobin A1c[HbA1c] > 8% or 64mmol/mol);
9. Treatment with immunosuppressants within 12 weeks prior to randomization, including but not limited to cyclophosphamide, azathioprine, mycophenolate, leflunomide, tacrolimus, cyclosporine, Tripterygium wilfordii;
10. Treatment with anti-CD20 therapy (for example, Rituximb Injection) within 24 weeks prior to randomization;
11. Received systemic glucocorticoid treatment within 12 weeks prior to randomization, excluding the followings: ① received systemic treatment with prednisolone ≤ 0.5mg/kg or equivalent glucocorticoid for non- IgA nephropathy for no more than 3 courses (≤ 2 weeks per course) in the past 52 weeks; ② topical administration or nasal inhalation;
12. Had hospitalization or intravenous anti-infective therapy for active infection within 4 weeks prior to randomization;
13. Patients with active tuberculosis;
14. Hepatitis B: patients with active or latent hepatitis B (potive HBcAb and HBV-DNA); According to the test results of hepatitis B five items, subjects with positive HBsAg will be excluded; subjects who are HBsAg-negative but HBcAb-positive, whether HBsAb is positive or negative, should be tested for HBV-DNA: if HBV-DNA is positive, patients should be excluded; if HBV-DNA is negative, patients can participate in the trial, and subjects are advised to take oral entecavir for prophylactic antiviral therapy during the trial;
15. Patients with hepatitis C;
16. Patients with HIV infection;
17. Patients with malignancy within the past 5 years, except for treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, colon polyps, or cervical cancer in situ;
18. Pregnant women, lactating women, and subjects with childbearing plans during the trial;
19. Allergic to biological products of human origin;
20. Participated in any clinical trial within 4 weeks or within 5 times the half-life of the investigational drug participating (whichever is longer) prior to randomization;
21. Received live vaccination within 4 weeks prior to randomization;
22. Drug or alcohol abuse/dependence within 52 weeks prior to randomization;
23. Other circumstances that, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in urine protein creatinine ratio (UPCR) | 39 weeks
  Based on a 24-hour urine collections.
Annualized estimated glomerular filtration rate (eGFR) slope | 104 weeks
  eGFR is calculated using the CKD-EPI formula.

SECONDARY OUTCOMES:
Proportion of patients with a 30% decrease in estimated glomerular filtration rate (eGFR) compared with baseline | 39 weeks
  eGFR is calculated using the CKD-EPI formula.
Time to 30% reduction from baseline in eGFR | up to 104 weeks
  eGFR is calculated using the CKD-EPI formula and confirmed by a second sample collection and calculation after at least 4 weeks.
Proportion of patients with a 40% decrease in estimated glomerular filtration rate (eGFR) compared with baseline | up to 104 weeks
  eGFR is calculated using the CKD-EPI formula and confirmed by a second sample collection and calculation after at least 4 weeks.
Proportion of patients received rescue treatment. | up to 104 weeks
  patients using systemic immunosuppressive medications, glucocorticoids (GCSs), etc.
Incidence and severity of adverse events | up to 104 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Change from baseline in urine protein creatinine ratio (UPCR) | 52 weeks,78 weeks,104 weeks
  Based on 24-hour urine collections.
Change from baseline in estimated glomerular filtration rate (eGFR) | 39 weeks, 52 weeks,78 weeks,104 weeks
  eGFR is calculated using the CKD-EPI formula.
Change from baseline in UACR in urine albumin-to-creatinine ratio (UACR) | 39 weeks, 52 weeks,78 weeks,104 weeks
  Based on 24-hour urine collections.
Time to composite endpoint event | up to 104 weeks
  The composite endpoint event is defined as initiation of maintenance renal dialysis (for at least 1 month), eGFR <15 mL/min/1.73 m^2, renal transplant, or death due to renal failure. eGFR is calculated using the CKD-EPI formula (CKD-EPI).
Proportion of patients achieving urine protein creatinine ratio (UPCR) < 0.8 g/g | 39 weeks, 52 weeks,78 weeks,104 weeks
  UPCR is calculated based on 24-hour urine collections;
Annualized estimated glomerular filtration rate (eGFR) slope | 52 weeks
  eGFR is calculated using the CKD-EPI formula.

OTHER OUTCOMES:
Change from baseline in 24-hour urine protein | 39 weeks
  based on 24-hour urine collections

CONTACTS AND LOCATIONS:
Overall Officials: Jicheng Lv, M.D., Principal Investigator — Peking University First Hospital
Locations (101):
- China (101):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The First Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Handan First Hospital, Handan, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theatre Command, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital，Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo Municipal Hospital of Traditional Chinese Medicine, Ningbo, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang
  - Tongde Hospital of Zhejing Province, Hangzhou, Zhejing

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639